CLINICAL TRIAL: NCT05157867
Title: In Vivo Effects of Amylase Trypsin Inhibitors From Wheat in the Human Gut: Proof of Cause of Non-coeliac Wheat Sensitivity in Irritable Bowel Syndrome?
Brief Title: In Vivo Effects of Amylase Trypsin Inhibitors
Acronym: ATI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL77666.608.21
Record Dates: First submitted 2021-10-06; First posted 2021-12-15 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Non-Coeliac Wheat Sensitivity (NCWS); Irritable Bowel Syndrome
Keywords: Non-Coeliac Wheat Sensitivity; Irritable Bowel Syndrome; Amylase Trypsin Inhibitors
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, cross-over study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amylase trypsin inhibitors (ATIs), then placebo (Experimental): Test day 1: intraduodenal administration of amylase trypsin inhibitors (ATIs) isolated from Triticum aestivum (bread wheat), dissolved in physiological saline. After a wash-out period of 4-6 weeks, test day 2: intraduodenal administration of placebo (physiological saline).
  Interventions: Other: Amylase trypsin inhibitors; Other: Placebo
- Placebo, then Amylase trypsin inhibitors (Experimental): Test day 1: intraduodenal administration of placebo (physiological saline). After a wash-out period of 4-6 weeks, test day 2: intraduodenal administration of amylase trypsin inhibitors (ATIs) isolated from Triticum aestivum (bread wheat), dissolved in physiological saline.
  Interventions: Other: Amylase trypsin inhibitors; Other: Placebo

INTERVENTIONS:
Other: Amylase trypsin inhibitors — Intraduodenal administration of amylase trypsin inhibitors (ATIs) isolated from Triticum aestivum (wheat), dissolved in physiological saline.
Other: Placebo — Intraduodenal administration of placebo (physiological saline).

SUMMARY:
Wheat is the most important staple food consumed in the Western world and provides beneficial health effects and functional properties. Nevertheless, an increasing proportion of the general population is avoiding or reducing its consumption of wheat products due to self-reported gastrointestinal (GI) symptoms, such as patients with non-coeliac wheat sensitivity (NCWS) and/or irritable bowel syndrome (IBS). There is increasing evidence that the amylase trypsin inhibitors (ATIs), accounting for up to 15% of wheat proteins, play a role in the symptom generation in NCWS and IBS. In vitro studies showed ATIs can induce an innate immune response via direct interaction with the toll-like receptor 4 (TLR4), activating the TLR4-MD2-CD14 complex with subsequent release of pro-inflammatory cytokines. These results were confirmed in mice. Furthermore, in mice ATIs triggered intestinal epithelial lymphocytosis and barrier dysfunction, and modified microbiota composition and metabolism. Thus far, there have been no placebo-controlled studies investigating these effects of isolated ATIs in human subjects. Understanding the role of ATIs in symptom generation in NCWS and IBS patients is important to provide these patients with appropriate dietary advice, improving their quality of life and decreasing their risk of nutritional deficiencies.

The investigators aim to perform a proof-of-concept study to assess the effect of ATIs on the intestinal barrier and immune function in healthy volunteers. The investigators hypothesise that the ATIs either directly affect the intestinal barrier function, or indirectly by activating an immune response via TLR4.

The study conforms a randomized, double-blind, placebo-controlled, cross-over design, using healthy human volunteers (male and female), 18-65 years old. Volunteers will each undergo two test days, separated by a wash-out period of at least 4 weeks. At the test day, volunteers receive either isolated ATIs or placebo (physiological saline), ingested using a nasogastric intraduodenal feeding catheter.

ELIGIBILITY:
Inclusion Criteria:

1. Based on medical history and previous self-admitted examination, no gastrointestinal complaints and/or disease can be defined.
2. Age between 18 and 65 years.
3. Body Mass Index (BMI) between 20 and 30 kg/m2.

Exclusion Criteria:

1. History of severe cardiovascular, respiratory, urogenital, gastrointestinal/hepatic, hematological/immunologic, HEENT (head, ears, eyes, nose, throat), dermatological/connective tissue, musculoskeletal, metabolic/nutritional, endocrine, neurological/psychiatric diseases, allergy, major surgery and/or laboratory assessments which might limit participation in or completion of the study protocol. The severity of the disease (major interference with the execution of the experiment or potential influence on the study outcomes) will be decided by the principal investigator.
2. Use of medication, including vitamin supplementation, pre- and probiotic supplementation, except oral contraceptives, within 14 days prior to testing.
3. Administration of investigational drugs or participation in any scientific intervention study, which may interfere with this study (to be decided by the principal investigator), in the 180 days prior to the study.
4. Major abdominal surgery interfering with gastrointestinal function (uncomplicated appendectomy, cholecystectomy and hysterectomy allowed, and other surgery upon judgement of the principal investigator).
5. Pregnancy, lactation.
6. Excessive alcohol consumption (> 14 alcoholic consumptions per week).
7. Smoking.
8. Drug use.
9. Blood donation within 3 months before or after the study period.
10. Self-admitted HIV-positive state.
11. Plan to lose weight or follow a specific diet (e.g. weight loss or gluten-free diet) within the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Difference in gene expression associated with intestinal barrier function, measured in duodenal biopsies collected after intervention with ATIs or placebo | Biopsies will be collected 2 hours after administration of ATIs or placebo, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Gene expression associated with intestinal barrier function, such as gene expression of tight junction and adherens junction proteins: e.g. peri-junctional Factin, myosin, ZO-1, claudin-3, occluding, myosin light chain kinase, phosphorylated myosin light chain, E-cadherin.
  Duodenal biopsies will be obtained using upper gastrointestinal endoscopy.

SECONDARY OUTCOMES:
Difference in protein levels associated with intestinal barrier function, measured in duodenal biopsies collected after intervention with ATIs or placebo. | Biopsies will be collected 2 hours after administration of ATIs or placebo, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Expression of proteins associated with intestinal barrier function, such as tight junction and adherens junction proteins by Western blot and immunofluorescent staining. Duodenal biopsies will be obtained using upper gastrointestinal endoscopy.
Differences in gene expression associated with immune function, measured in duodenal biopsies collected after intervention with ATIs or placebo. | Biopsies will be collected 2 hours after administration of ATIs or placebo, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Gene expression associated with immune activation, such as TLR4, and pro-inflammatory cytokines and antimicrobiota peptides.
  Duodenal biopsies will be obtained using upper gastrointestinal endoscopy.
Differences in infiltration of immune cells in duodenal tissue, measured in duodenal biopsies collected after intervention with ATIs or placebo. | Biopsies will be collected 2 hours after administration of ATIs or placebo, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Infiltration of immune cells (neutrophils, mast cells, dendritic cells) into duodenal tissue by immunofluorescent staining. Duodenal biopsies will be obtained using upper gastrointestinal endoscopy.
Difference in change in gastrointestinal symptoms from baseline after intervention with ATIs or placebo. | Various time points throughout each test day: 1 hour before and 5 minutes before intervention with ATIs or placebo, and 1 hour, 2 hours and 12 hours after intervention with ATIs or placebo
  Measured on the Visual Analogue Scale ranged from 0-100, in which 0 is absence of symptoms and 100 is severe symptoms; ATIs vs placebo
Difference in blood immune cell populations after intervention with ATIs or placebo | Blood samples will be collected directly after upper gastrointestinal endoscopy, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Quantification of immune cell populations (T helper cells, cytotoxic T cells, CD25+ effector T cells, CD69+ effector T cells, regulatory T cells, and NK-cells) in whole blood.
Difference in blood biomarkers of immune stimulation after intervention with ATIs or placebo | Blood samples will be collected directly after upper gastrointestinal endoscopy, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Measurement of biomarkers of immune stimulation (such as the human cytokines IL-10, TGF-β, IL-12p40 subunit, IL-12p70 subunit, IL-1β, IL-2, IL-6, IL-4, IL-17, IL-22 and IFN-γ, TNFα) in whole blood.
Blood markers for intestinal barrier function after intervention with ATIs or placebo | Blood samples will be collected directly after upper gastrointestinal endoscopy, on two separate test days. The test days are separated by a wash-out period of 4-6 weeks.
  Markers for intestinal barrier function (plasma citrulin, metabolites) and small intestinal mucosal tissue injury (intestinal fatty acid binding protein (I-FABP)), measured in whole blood.

OTHER OUTCOMES:
Participant characteristics | Data on demographic factors and medical history will be collected during the screening visit
  To assess suitability for participation of to characterise the study population, data will be collected on demographics and medical history using screening questionnaires.
One-day food record to ensure dietary intake is similar during the 24 hours before testday 1 and testday 2. | 24 hours prior to testday 1, and after a wash-out period of 4-6 weeks, also during the 24 hours prior to testday 2
  Participants will be asked to repeat intake prior to testday 1 on the day prior to testday 2. Thus, the intake is written down during the 24 hours prior to test day 1, and repeated (and again written down) during the 24 hours prior to testday 1, which is 4-6 weeks after test day 1.

CONTACTS AND LOCATIONS:
Overall Officials: Daisy MAE Jonkers, Prof, PhD, Principal Investigator — Maastricht University

IPD SHARING:
Plan to Share IPD: No